CLINICAL TRIAL: NCT01989637
Title: Effects of a Freeze Dried Strawberry Powder on Postprandial Vascular Function and Blood Markers of Cardiovascular Risk
Brief Title: Effect of Strawberries on Cardiovascular Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PKE STR
Record Dates: First submitted 2013-07-31; First posted 2013-11-21 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strawberry Meal (Experimental): 40 g freeze-dried strawberries included in test meal
  Interventions: Dietary Supplement: Strawberry Meal
- Control Meal (Placebo Comparator): Control consisting of matched test meal with strawberry flavoring instead of freeze-dried strawberry powder
  Interventions: Dietary Supplement: Control Meal

INTERVENTIONS:
Dietary Supplement: Strawberry Meal — High-fat meal (50 g total fat) with 40 g freeze dried strawberry powder
  Arms: Strawberry Meal
Dietary Supplement: Control Meal — High-fat meal (50 g total fat) with a matched placebo powder containing no strawberry bioactives
  Arms: Control Meal

SUMMARY:
It is important to identify and evaluate foods, such as strawberries, that can improve established and emerging cardiovascular risk factors, such as postprandial lipid and glycemic responses, and vascular health. Postprandial derangements may affect multiple metabolic pathways that lead to increased arterial stiffness. Research has demonstrated the potential of strawberries to ameliorate postprandial responses to a high fat/high glucose meal. Further research is needed to demonstrate this effect in better controlled clinical studies and explore whether metabolic effects lead to improved arterial health.

The investigators propose to examine the effects of adding 40 g of freeze-dried strawberry powder to a high fat/high glucose meal on postprandial cardiovascular risk factor including lipids, insulin, glucose, and arterial stiffness and central blood pressure. The investigators hypothesize that the bioactive components of strawberry powder will attenuate postprandial lipemic and glycemic responses, as well as improve measures of arterial health.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years of age
* LDL-C below 160 mg/dL
* Triglycerides below 350 mg/dL
* No stage II hypertension (BP below 160/100 mmHg)
* Not taking medication for elevated lipids, blood pressure, or glucose

Exclusion Criteria:

* Allergies to strawberries
* Known intolerance to high fat meals
* History of cardiovascular disease, kidney disease, diabetes or inflammatory diseases such as GI disorders and arthritis
* Use of non-steroidal anti-inflammatory or immunosuppressant drugs
* Conditions requiring the use of steroids
* Use of medication or supplements for elevated lipids, blood pressure or glucose

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postprandial central blood pressure and arterial stiffness | 2 and 4 hours

SECONDARY OUTCOMES:
Postprandial changes in insulin | 0, 0.5, 1, 2, and 4 hours
Postprandial changes in glucose | 0, 0.5, 1, 2, and 4 hours
Postprandial changes in markers of inflammation/oxidative stress | 0, 0.5, 1, 2, and 4 hours
Change from baseline in postprandial triglycerides at 0.5, 1, 2, and 4 hours | 0.5, 1, 2, and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Penny M Kris-Etherton, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Burdge GC, Calder PC. Plasma cytokine response during the postprandial period: a potential causal process in vascular disease? Br J Nutr. 2005 Jan;93(1):3-9. doi: 10.1079/bjn20041282. PMID 15705218
- [Background] Jennings A, Welch AA, Fairweather-Tait SJ, Kay C, Minihane AM, Chowienczyk P, Jiang B, Cecelja M, Spector T, Macgregor A, Cassidy A. Higher anthocyanin intake is associated with lower arterial stiffness and central blood pressure in women. Am J Clin Nutr. 2012 Oct;96(4):781-8. doi: 10.3945/ajcn.112.042036. Epub 2012 Aug 22. PMID 22914551
- [Background] Erlund I, Koli R, Alfthan G, Marniemi J, Puukka P, Mustonen P, Mattila P, Jula A. Favorable effects of berry consumption on platelet function, blood pressure, and HDL cholesterol. Am J Clin Nutr. 2008 Feb;87(2):323-31. doi: 10.1093/ajcn/87.2.323. PMID 18258621
- [Background] Basu A, Fu DX, Wilkinson M, Simmons B, Wu M, Betts NM, Du M, Lyons TJ. Strawberries decrease atherosclerotic markers in subjects with metabolic syndrome. Nutr Res. 2010 Jul;30(7):462-9. doi: 10.1016/j.nutres.2010.06.016. PMID 20797478
- [Background] Basu A, Wilkinson M, Penugonda K, Simmons B, Betts NM, Lyons TJ. Freeze-dried strawberry powder improves lipid profile and lipid peroxidation in women with metabolic syndrome: baseline and post intervention effects. Nutr J. 2009 Sep 28;8:43. doi: 10.1186/1475-2891-8-43. PMID 19785767
- [Background] Burton-Freeman B, Linares A, Hyson D, Kappagoda T. Strawberry modulates LDL oxidation and postprandial lipemia in response to high-fat meal in overweight hyperlipidemic men and women. J Am Coll Nutr. 2010 Feb;29(1):46-54. doi: 10.1080/07315724.2010.10719816. PMID 20595645
- [Background] Jenkins DJ, Nguyen TH, Kendall CW, Faulkner DA, Bashyam B, Kim IJ, Ireland C, Patel D, Vidgen E, Josse AR, Sesso HD, Burton-Freeman B, Josse RG, Leiter LA, Singer W. The effect of strawberries in a cholesterol-lowering dietary portfolio. Metabolism. 2008 Dec;57(12):1636-44. doi: 10.1016/j.metabol.2008.07.018. PMID 19013285
- [Background] Zunino SJ, Parelman MA, Freytag TL, Stephensen CB, Kelley DS, Mackey BE, Woodhouse LR, Bonnel EL. Effects of dietary strawberry powder on blood lipids and inflammatory markers in obese human subjects. Br J Nutr. 2012 Sep;108(5):900-9. doi: 10.1017/S0007114511006027. Epub 2011 Nov 9. PMID 22068016
- [Background] Skulas-Ray AC, Kris-Etherton PM, Teeter DL, Chen CY, Vanden Heuvel JP, West SG. A high antioxidant spice blend attenuates postprandial insulin and triglyceride responses and increases some plasma measures of antioxidant activity in healthy, overweight men. J Nutr. 2011 Aug;141(8):1451-7. doi: 10.3945/jn.111.138966. Epub 2011 Jun 22. PMID 21697300
- [Background] de la Garza AL, Milagro FI, Boque N, Campion J, Martinez JA. Natural inhibitors of pancreatic lipase as new players in obesity treatment. Planta Med. 2011 May;77(8):773-85. doi: 10.1055/s-0030-1270924. Epub 2011 Mar 16. PMID 21412692
- [Derived] Richter CK, Skulas-Ray AC, Gaugler TL, Lambert JD, Proctor DN, Kris-Etherton PM. Incorporating freeze-dried strawberry powder into a high-fat meal does not alter postprandial vascular function or blood markers of cardiovascular disease risk: a randomized controlled trial. Am J Clin Nutr. 2017 Feb;105(2):313-322. doi: 10.3945/ajcn.116.141804. Epub 2016 Dec 21. PMID 28003205